CLINICAL TRIAL: NCT05793216
Title: VestibulOTherapy: Vestibular Impact on Learning
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: VestibulOTherapy (Industry)
Collaborators: University of Wisconsin, La Crosse (Other); Boston University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 03072023
Record Dates: First submitted 2023-03-08; First posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Vestibular Disorder; Educational Problems; Attention Deficit Disorder
Keywords: vestibular; occupational therapy; children; educational outcomes
MeSH Terms: conditions — Vestibular Diseases; Attention Deficit Disorder with Hyperactivity | interventions — Occupational Therapy

STUDY DESIGN:
Intervention Model Description: This program involves a multiple baseline design for a group of students ages 6-9 years. The intervention will last for 8 weeks with educational outcomes monitored before, during, and after the intervention. With final reporting at 6 months post intervention.
Masking Description: Outcome measures will be reviewed by a neutral party to avoid bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Classroom interventions (Experimental): Students within five classrooms will engage in prescribed vestibular activities embedded within learning curricula to determine the impact of the intervention on learning outcomes, particularly memory, sequencing, attention, and ordinance related outcomes.
  Interventions: Behavioral: VestibulOTherapy

INTERVENTIONS:
Behavioral: VestibulOTherapy — For this study, the following activity-orientated interventions will occur within the natural learning environments so that generous opportunities exist for neural plasticity and growth.
  Each student will be engaged in 20-30 minutes/day of intermittent classroom activities, plus 20-30- minutes of daily stability work embedded into classroom routines including stabilizing self on a Hokki stool or t-stool or standing on a balance board during sedentary work, such as circle time or read-a-loud.
  Other Names: occupational therapy

SUMMARY:
Research Question: Will daily engagement in activities tailored to the evidence-based vestibular research result in improved attention and learning outcomes for children ages 6-9 years of age after an 8-week classroom-based intervention?

DETAILED DESCRIPTION:
"Vestibulotherapy" is an emerging frame of reference aiming to help neurotypical children with under-performing vestibular systems develop neural pathways supporting communication and learning.

Theory based upon systematic review: Given adequate vestibular activation through targeted activities (in an otherwise under-performing vestibular system), myelination and neuroplasticity propagate along learning pathways leading to greater neural connectivity and efficiency for sequencing, ordinance, attention, memory, body schema, spatial cognition, executive function, and interoception.

As a result of prescribed vestibular interventions and gained attributes supporting learning, students will experience increased academic growth and success as outlined by the following model.

ELIGIBILITY:
Inclusion Criteria:

* neurotypical development
* between the ages of 6-10 years of age
* performance challenges in school in the areas of math, spelling, organization, sequencing, attention, or engagement
* demonstrate attributes of vestibular dysfunction per the Vestibular Profile
* may have ADD or ADHD
* May have challenges with speech articulation
* good potential for learning and engaging in prescribed interventions

Exclusion Criteria:

* Neurodiverse development (with the exception of ADHD or ADD)
* Absence of vestibular challenges
* Absence of learning challenges.
* unable to participate in interventions on a routine basis due to attendance or other limitations.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Estimated)
Dates: Start 2023-03-07 (Actual); Primary Completion 2023-05-05 (Estimated); Study Completion 2023-10-25 (Estimated)

PRIMARY OUTCOMES:
Change in Academic Score reporting | Baseline data established at recruitment, followed by weekly data collection of scores from spelling and math for twelve weeks, and again once at three-months post intervention
  Academic record review: Math, spelling, and reading records from the 1st Semester of school will indicate trends in student performance. Immediately following and six months post-intervention, the trends will be compared to determine if a significant change occurs in these dependent variables. During and immediately following the intervention, spelling and math tests will be taken on consistent days of the week to avoid variabilities in data. Numerical data will be graphed to illustrate and examine trends and slope over time to determine significance of change.
Vestibular Attributes | up to twelve weeks
  Vestibular Profile - Pediatric (VP-P) will be completed at recruitment. The most salient attributes will be monitored weekly throughout the intervention.
Time on Task / Attention | up to twelve weeks
  Time on Task measures reflecting active participation and attention during instruction

CONTACTS AND LOCATIONS:
Overall Officials: Constance L Wall, OTD, Principal Investigator — Boston University
Locations (1):
- School District of La Crosse, La Crosse, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification will be shared through publications related to research outcomes.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Immediately following publication. No end date.
Access Criteria: Anyone who wishes to access the data.

REFERENCES:
- [Background] Besnard S, Tighilet B, Chabbert C, Hitier M, Toulouse J, Le Gall A, Machado ML, Smith PF. The balance of sleep: Role of the vestibular sensory system. Sleep Med Rev. 2018 Dec;42:220-228. doi: 10.1016/j.smrv.2018.09.001. Epub 2018 Sep 8. PMID 30293919
- [Background] Hitier M, Besnard S, Smith PF. Vestibular pathways involved in cognition. Front Integr Neurosci. 2014 Jul 23;8:59. doi: 10.3389/fnint.2014.00059. eCollection 2014. PMID 25100954
- [Background] Emami Kashfi T, Sohrabi M, Saberi Kakhki A, Mashhadi A, Jabbari Nooghabi M. Effects of a Motor Intervention Program on Motor Skills and Executive Functions in Children With Learning Disabilities. Percept Mot Skills. 2019 Jun;126(3):477-498. doi: 10.1177/0031512519836811. Epub 2019 Mar 16. PMID 30879395
- [Background] Lopez C, Toupet M, van Nechel C, Bozorg Grayeli A. Editorial: Role of Inner Ear in Self and Environment Perception. Front Neurol. 2020 Feb 20;11:22. doi: 10.3389/fneur.2020.00022. eCollection 2020. No abstract available. PMID 32153485
- [Background] Lotfi Y, Rezazadeh N, Moossavi A, Haghgoo HA, Rostami R, Bakhshi E, Badfar F, Farokhi Moghadam S, Sadeghi-Firoozabadi V, Khodabandelou Y. Rotational and Collic Vestibular-Evoked Myogenic Potential Testing in Normal Developing Children and Children With Combined Attention Deficit/Hyperactivity Disorder. Ear Hear. 2017 Nov/Dec;38(6):e352-e358. doi: 10.1097/AUD.0000000000000451. PMID 28562425
- [Background] Mast FW, Preuss N, Hartmann M, Grabherr L. Spatial cognition, body representation and affective processes: the role of vestibular information beyond ocular reflexes and control of posture. Front Integr Neurosci. 2014 May 27;8:44. doi: 10.3389/fnint.2014.00044. eCollection 2014. PMID 24904327
- [Background] Matuszkiewicz M, Galkowski T. Developmental Language Disorder and Uninhibited Primitive Reflexes in Young Children. J Speech Lang Hear Res. 2021 Mar 17;64(3):935-948. doi: 10.1044/2020_JSLHR-19-00423. Epub 2021 Feb 23. PMID 33621124
- [Background] Melo RS, Lemos A, Paiva GS, Ithamar L, Lima MC, Eickmann SH, Ferraz KM, Belian RB. Vestibular rehabilitation exercises programs to improve the postural control, balance and gait of children with sensorineural hearing loss: A systematic review. Int J Pediatr Otorhinolaryngol. 2019 Dec;127:109650. doi: 10.1016/j.ijporl.2019.109650. Epub 2019 Aug 21. PMID 31466025